CLINICAL TRIAL: NCT04204629
Title: A Randomized, Open-label, Single Dose, Crossover Study to Investigate the Effect of Food on the Pharmacokinetics and Pharmacodynamics of HIP1601 40 mg in Healthy Volunteers
Brief Title: Food-effect on PK and PD of Single Oral Dose of HIP1601 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ESOM-103
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1: Fasted state + HIP1601 Period 2: Fed state + HIP1601
  Interventions: Drug: HIP1601 40mg
- Sequence 2 (Experimental): Period 1: Fed state + HIP1601 Period 2: Fasted state + HIP1601
  Interventions: Drug: HIP1601 40mg

INTERVENTIONS:
Drug: HIP1601 40mg — Single dosing of HIP1601 40mg, PO
  Other Names: HIP1601

SUMMARY:
Primary objective - To evaluate food effect on the pharmacokinetics and the pharmacodynamics (PD) of a single oral dose of HIP1601 in healthy subjects under fed or fasting condition.

Secondary objectives

- To evaluate the safety of single oral dose of HIP1601 in healthy subjects under fed or fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female healthy volunteers in the age between 19 and 50 years old.
* Body mass index (BMI) in the range of 19 to 28 kg/m2 and weight 55.0kg to 90.0kg.
* Helicobacter pylori (H. Pylori) negative.
* After fully hearing and understanding the details of this clinical trial, Subjects who have willingness to sign of informed consent before the screening.
* Subject who are eligible from physical examination, clinical laboratory test by investigators judgment.

Exclusion Criteria:

* Gastrointestinal disorders (gastrointestinal ulcers, gastritis, stomach cramps, gastro-esophageal reflux disease, Crohn's disease or chronic pancreatitis) or gastrointestinal surgery (except for simple cecal or hernia surgery) which may affect the safety and pharmacokinetic evaluation of test drug.
* Subjects who have a history of hypersensitivity or clinically significant hypersensitivity to esomeprazole or the same component or other drugs (aspirin, antibiotics, etc.).
* Blood serum aspartate aminotransferase and alanine aminotransferase exceed 1.5 times the upper limit of normal range from screening laboratory results before randomization.
* Subject who continues to drink (21 units / week, 1 unit = 10 g of pure alcohol) within a month before the screening visit or who cannot abstain during the hospital stay.
* Heavy smoker (>10 cigarettes/day).

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Cmax | Blood sampling during 24 hours after administration
  Maximum observed concentration after dose
Area Under the plasma concentration versus time Curve(AUC)last | Blood sampling during 24 hours after administration
  Area under the plasma concentration versus time curve from dosing to the last quantifiable concentration
Integrated gastric acidity for 24-hour | Blood sampling during 24 hours after administration
  Percent decrease from baseline in integrated gastric acidity for 24-hour interval after dose

SECONDARY OUTCOMES:
Tmax | Blood sampling during 24 hours after administration
  Time of Cmax over the time span specified
AUCinf | Blood sampling during 24 hours after administration
  Area under the plasma concentration versus time curve from the time of dosing to time extrapolated to infinitely
t1/2 | Blood sampling during 24 hours after administration
  Terminal half-life
Clearance/F | Blood sampling during 24 hours after administration
  Apparent total body clearance after extravascular administration, calculated as Dose/AUCinf
Vd/F | Blood sampling during 24 hours after administration
  Apparent volume of distribution after extravascular administration, calculated as Dose/(λzㆍAUCinf)
Duration of time intra-gastric pH 4.0 or higher | Blood sampling during 24 hours after administration
  Percent of time with intra-gastric pH greater than 4.0 for 24-hour interval after dose
Median pH | Blood sampling during 24 hours after administration
  Median intra-gastric pH for 24-hour interval after dose

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, Principal Investigator — Seoul National University Hospital, Seoul, Korea
Locations (1):
- Seoul National University Biomedical Research Institute, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No